CLINICAL TRIAL: NCT01260025
Title: Dose Escalation Study of Tolerability and Pharmacokinetics of PEDylated Recombinant Human Endostatin(M2ES)in the Treatment of Advanced Solid Tumor
Brief Title: Tolerability and Pharmacokinetics of M2ES in the Treatment of Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009L01132
Record Dates: First submitted 2010-09-08; First posted 2010-12-15 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Tolerability; Pharmacokinetics; Endostatin
Keywords: Tolerability; Pharmacokinetics; Endostatin; antiangiogenesis; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEDylated Recombinant Human Endostatin (Experimental): PEDylated Recombinant Human Endostatin
  Interventions: Drug: PEDylated Recombinant Human Endostatin

INTERVENTIONS:
Drug: PEDylated Recombinant Human Endostatin — The initial dose of PEDylated Recombinant Human Endostatin (M2ES) will be 7.5mg/m2.Dose Escalation to a next higher level will occur when 3 patients in the same dose level complete 28 days of continuous treatment without experiencing a dose-limiting toxicity.
  Other Names: M2ES

SUMMARY:
1. MTD and DLT of M2ES
2. Pharmacokinetics of M2ES

DETAILED DESCRIPTION:
Patients received infusion of M2ES for 120 minutes weekly（d1,d8,d15）by calculated pump and underwent evaluation of vital signs including blood pressure, pulse, respiratory rate, and temperature before treatment, at intervals during infusion, and hourly for 6 hours after infusion. After infusion, patients underwent serial pharmacokinetic sampling. All patients were seen weekly during the study therapy and follow-up and underwent evaluation with physical examination including ECOG performance status, vital signs, and laboratory evaluation with complete blood count with manual differential, chemistry evaluation, prothrombin time/partial thromboplastin time, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;Genders eligible for study: both;
* Histologic diagnosis of solid malignancies ;
* Performance status of 0 or 1;
* Tumor not amenable to standard curative or palliative therapy;
* life expectancy beyond 3 months;
* Ability to give signed informed consent

Exclusion Criteria:

* Pregnancy or lactation;
* Had a history of brain metastasis or a primary brain tumor;
* An active, potentially severe autoimmune disease;
* Serum creatinine ≥1.5mg/dl or a calculated creatinine clearance <60ml/min; WBC count < 2.0×109/L，hemoglobin < 90g/L，and platelet count < 100×109/L; Total bilirubin value < 2.0 times the upper limit of normal (ULN), ALT level < 2.0 times ULN, AST < 2.0 times ULN;
* Positive of anti-HIV antibodies;
* An active infection;
* had received chemotherapy or immunotherapy within the prior 4 weeks before study entry
* Participation in a clinical study during the last 28 days
* QTc with Bazett's correction unmeasurable or ≥ 480 msec on screening ECG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maxinum tolerated dose of M2ES | one month
  To assess the adverse events

SECONDARY OUTCOMES:
Tumor response rate | one month
  To assess the tumor response rate of M2ES in patients with solid, malignant tumours
Pharmacokinetic effect | one month
  Pharmacokinetic effect of M2ES in patients with solid, malignant tumours
DLT of M2ES | one month
  To assess the adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China